CLINICAL TRIAL: NCT07362433
Title: The BLAAAST Trial: Bangladesh Lung Auscultation AI for Antibiotic Stewardship Randomized Controlled Trial
Brief Title: Trial of an AI-enabled Digital Stethoscope to Improve Antibiotic Stewardship
Acronym: BLAAAST
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Projahnmo Research Foundation (Other); University College, London (Other); Thomas Jefferson University (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: IRB00451423; R01HD115597 (NIH)
Record Dates: First submitted 2026-01-21; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Infections in Children
Keywords: Digital auscultation; Automated digital stethoscope; Artificial intelligence lung sound analysis; Pediatric pneumonia; Integrated Management of Childhood Illness (IMCI); Antibiotic stewardship; Point-of-care respiratory diagnostics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IMCI guidelines enhanced by automated digital stethoscope (Experimental): IMCI child pneumonia guideline care enhanced by a commercially available automated digital stethoscope.
  Interventions: Device: Automated digital stethoscope
- IMCI guidelines without automated digital stethoscope enhancement (No Intervention): Standard IMCI child pneumonia care that is not enhanced by a commercially available automated digital stethoscope.

INTERVENTIONS:
Device: Automated digital stethoscope — The digital auscultation system intervention is comprised of a wireless electronic stethoscope and mobile phone application that records and analyzes lung sounds using an automated algorithm. The system has achieved European Union Class IIa medical device certification (EU Class IIa), which confirms its safety and clinical performance, and permits its use in clinical facilities by healthcare workers.
  Arms: IMCI guidelines enhanced by automated digital stethoscope

SUMMARY:
Antibiotics are a mainstay of the treatment of lower respiratory infections in young children even though most episodes are caused by self-limiting viruses. Innovative child friendly tools that improve the diagnosis of respiratory illnesses, safely reduce the unnecessary use of antibiotics, and are suitable for implementation in resource-constrained settings are urgently required to safely improve antibiotic stewardship and stem the rising rates of antibiotic resistance globally.

In the Bangladesh Lung Auscultation Artificial Intelligence for Antibiotic Stewardship Trial (BLAAAST) the investigators aim to determine whether treatment failure frequency among children in rural Bangladesh managed by clinical guidelines enhanced by a commercially available, artificial intelligence (AI)-enabled digital stethoscope is non-inferior to guidelines alone. The investigators hypothesize treatment failure frequency among 'enhanced IMCI' participants will be no worse than standard care by a +/-2% margin, safely reducing antibiotic use by 50-60%. The investigators will also evaluate if a diagnostic strategy enhanced by an AI-enabled digital stethoscope is a sustainable alternative to standard care for children in rural Bangladesh. The investigators hypothesize that care augmented by an AI-enabled digital stethoscope will have additional benefits via reduced antibiotic use that will outweigh digital auscultation costs resulting in cost-effectiveness compared to current practice.

BLAAAST affords a unique opportunity to evaluate the efficacy of clinical guidelines enhanced by an AI-enabled digital stethoscope on child pneumonia outcomes in Bangladesh, if digital auscultation may be instrumental in the wider antibiotic stewardship strategy, and whether a digital stethoscope diagnostic tool is cost-effective in the care of children with respiratory illnesses.

DETAILED DESCRIPTION:
Participants will be screened for eligibility by study physicians. Children who screen positive will then be assessed for eligibility. Written informed consent will be obtained. All enrolled children will have a lung sound recording obtained. Study physicians will sequentially record lung sounds using the digital stethoscope from four chest positions (two anterior and two posterior) on participants. Each chest position recording is 15 seconds, and the overall procedure ~2 minutes. Lung sound recordings will be transferred to an encrypted tablet and analyzed by the convolutional neural network model to automatically detect normal and abnormal lung sounds. Blocked randomization will occur after the recording has been completed. Children who consent and meet eligibility criteria will be randomized into one of two arms.

Children randomized to the intervention will receive amoxicillin syrup (250mg/5ml concentration) or placebo based on the automated algorithm's lung sound classification. Children receiving a positive digital stethoscope result will receive amoxicillin while children receiving a negative digital stethoscope results will receive placebo. All children in the control arm (standard care) will receive amoxicillin. Treatment duration will be five days per Integrate Management of Childhood Illnesses (IMCI) guidelines, administering the study product twice daily. Children randomized to the control group will receive amoxicillin syrup (250mg/5ml concentration) for five days as all controls will meet IMCI pneumonia criteria. Study physicians and caregivers in the IMCI clinic will be masked to the randomization group. Masking will be achieved by applying the digital stethoscope to all enrolled children and concealing the automated algorithm result on the device.

Trained community healthcare worker paramedics equipped a pulse oximeter and paracetamol will conduct home visits for all participants on study days 2, 3, 5, and 14 after enrollment (defined as Day 1). A study physician will conduct the day 7 study visit and assign the primary outcome. A 24-hour window period will be permitted for each home visit in the event that the participant is not available on the scheduled visit day.

Any child that meets treatment failure criteria will be immediately transported to the study facility (Upazila Health Complex) for study physician confirmation and further treatment planning. Similarly, an oxygen saturation measured as 90-94% will prompt referral to the study physician for assessment for treatment failure. Study physician confirmation is required for a treatment failure outcome. Caregivers will be provided a trial telephone hotline for communications between scheduled visits (by text message or phone call), should parental concerns arise between household visits. If caregivers prefer, the caregiver may also return to the study clinic for a study physician reassessment between community health worker (CHW) household visits.

For any participant receiving amoxicillin or placebo who is confirmed to have a World Health Organization (WHO)-defined emergency sign, WHO-defined clinical danger sign, or WHO-defined hypoxemia, and the child will be hospitalized and receive parenteral antibiotics according to WHO-guidelines and aligned with Bangladesh national guidelines. Further treatment and clinical management will be at the discretion of the treating physician. For any participant on amoxicillin or placebo who is confirmed to have lower chest wall indrawing and/or very fast breathing for age on day 7 and who is confirmed to be without any WHO-defined emergency signs, to be without any WHO-defined clinical danger signs, and to be without WHO-defined hypoxemia, then the child will be initiated on oral amoxicillin-clavulanic acid over a minimum of 5 days. Further treatment and clinical management will be at the discretion of the treating physician. Unblinding will occur only when knowledge of treatment allocation is essential for the clinical management of a participant or when required to address a serious adverse event or unexpected problem posing risk to participant safety.

Participants will be enrolled into the trial for a period of 2 weeks each. There is a minimum of 6 study visits. The use of a placebo in this study is justified to maintain participant adherence to the assigned treatment and ensure comparability between the intervention and control groups. Without a placebo, participants who do not receive antibiotics are likely to be dissatisfied and seek treatment from another provider, thereby introducing a protocol violation, observer bias, and compromising the study's validity by leading to an over- or underestimation of the true treatment effect. By ensuring blinding, the placebo is also crucial for reducing bias in outcome assessment by study investigators. In sum, by using a placebo, the study can accurately differentiate between the effects of appropriately withholding antibiotics and any potential treatment effects, thereby providing robust and reliable results that are most likely to impact on health policy.

With a sample size of 2500 and one-week (7 day) treatment failure rate in the placebo arm of the trial to be approximately 4% based on prior data, and the margin of non-inferiority was chosen to be 2% based on the largest clinically acceptable difference between treatment failure of the intervention compared to the standard care. Given these parameters, the investigators will have at least 80% power to reject the null hypothesis of inferiority given that the treatment failure rate in the intervention arm is equal to the placebo arm, at 4%, assuming a one-sided type one error of 0.05.

Requiring medical care, requiring hospitalization, and mortality among study participants will be recorded by the study as the 3 primary markers of safety. In addition to these 3 parameters, the investigators will collect data on all unexpected adverse events (AEs) that occur during the study period. AEs will be actively collected from enrollment through Day 14 post-enrollment, or until completion of all follow-up procedures, whichever occurs later.

Rigorous safety measures will be in place including eligibility restrictions to 'low risk' children with non-severe clinical pneumonia, a hotline for 24/7 communication, close household follow-up (at least 5 household visits, including daily over the first 3 days of illness), and facilitating participant clinic transportation if needed. The trial will have a Data Safety and Monitoring Board (DSMB) and Technical Advisory Group. If unscheduled healthcare facility visits are necessary, then participants will be reimbursed for any travel expenses incurred. Participants will not be directly compensated for study visits conducted in the home and for study visits coordinated with routine healthcare visits at hospitals.

ELIGIBILITY:
Inclusion Criteria:

* 2 to 59 months of age (60 days to 59 months 29 days),
* illness duration 14 days or less,
* meeting non-severe pneumonia criteria, and
* from the trial catchment areas.

Exclusion Criteria:

* prior participation,
* age <2 months or >59 months,
* illness duration >14 days,
* not meeting IMCI-defined non-severe pneumonia criteria,
* oxygen saturation (SpO2) <90%,
* moderate or severe malnutrition,
* known chronic disease,
* history of prematurity,
* one or more high risk clinical signs (any WHO-defined clinical danger sign and/or WHO-defined emergency sign),
* known antibiotic exposure in the past 1 week,
* non-respiratory illness requiring systemic antibiotic treatment according to IMCI guidelines.

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2500 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | 7 days
  Treatment failure (primary outcome) is defined as (1) death at any time on or before day 7, or (2) clinical deterioration (development of any WHO danger sign and/or any WHO emergency sign (i.e., 'high-risk' signs)) at any time on or before day 7, or (3) the presence of chest indrawing and/or very fast breathing for age on day 7 (not before day 7), or (4) lost-to-follow-up at any time on or before day 7, or (5) hospitalization for any reason at any time on or before day 7, or (6) a change in antibiotic treatment at any time on or before day 7. Clinical deterioration is defined as the development of (1) any WHO-defined clinical danger sign, and/or (2) WHO-defined emergency sign, and/or (3) hypoxemia (SpO2 <90%) at any time after enrollment.

SECONDARY OUTCOMES:
Treatment failure (modified) | 7 days
  Treatment failure (modified - secondary outcome) is defined as (1) death at any time on or before day 7, or (2) clinical deterioration (development of any WHO danger sign and/or any WHO emergency sign (i.e., 'high-risk' signs)) at any time on or before day 7, or (3) the presence of chest indrawing and/or fast breathing for age on day 7 (not before day 7), or (4) lost-to-follow-up at any time on or before day 7, or (5) hospitalization for any reason at any time on or before day 7, or (6) a change in antibiotic treatment at any time on or before day 7. Clinical deterioration is defined as the development of (1) any WHO-defined clinical danger sign, and/or (2) WHO-defined emergency sign, and/or (3) hypoxemia (SpO2 <90%) at any time after enrollment.
Treatment relapse | 14 days
  Treatment relapse (secondary outcome) is defined as (1) death at any time after day 7, or (2) clinical deterioration (development of any WHO danger sign and/or any WHO emergency sign (i.e., 'high-risk' signs)) at any time after day 7, or (3) the presence of chest indrawing and/or very fast breathing for age after day 7, or (4) hospitalization for any reason at any time after day 7. Clinical deterioration is defined as the development of (1) any WHO-defined clinical danger sign, and/or (2) WHO-defined emergency sign, and/or (3) hypoxemia (SpO2 <90%) at any time after day 7.
Subgroup analysis: Treatment failure stratified by age | 7 days
  Analysis of treatment failure (primary outcome definition) stratified by age
Subgroup analysis: Treatment failure stratified by sex | 7 days
  Analysis of treatment failure (primary outcome definition) stratified by sex
Subgroup analysis: Treatment failure stratified by study site | 7 days
  Analysis of treatment failure (primary outcome definition) stratified by study site
Digital stethoscope classification agreement | 1 day
  Among a subgroup of participants, the agreement between the digital stethoscope automated analysis classification and an expert review panel classification of lung sounds collected at enrollment.
Time to treatment failure in days | 7 days
  All treatment failure times in days, comparing the time until treatment failure between arms
Subgroup analysis: Treatment failure (modified definition) stratified by age | 7 days
  Analysis of treatment failure (modified definition) stratified by age
Subgroup analysis: Treatment relapse stratified by age | 14 days
  Analysis of treatment relapse stratified by age
Subgroup analysis: Treatment failure (modified definition) stratified by sex | 7 days
  Analysis of treatment failure (modified definition) stratified by sex
Subgroup analysis: Treatment relapse stratified by sex | 14 days
  Analysis of treatment relapse stratified by sex
Subgroup analysis: Treatment failure (modified definition) stratified by study site | 7 days
  Analysis of treatment failure (modified definition) stratified by study site
Subgroup analysis: Treatment relapse stratified by study site | 14 days
  Analysis of treatment relapse stratified by study site
Digital stethoscope sensitivity | 14 days
  Among a subgroup of participants, the sensitivity of the digital stethoscope diagnosis relative to a gold standard diagnosis assigned by expert review.
Digital stethoscope specificity | 14 days
  Among a subgroup of participants, the specificity of the digital stethoscope diagnosis relative to a gold standard diagnosis assigned by expert review.
Digital stethoscope positive predictive value | 14 days
  Among a subgroup of participants, the positive predictive value of the digital stethoscope diagnosis relative to a gold standard diagnosis assigned by expert review.
Digital stethoscope negative predictive value | 14 days
  Among a subgroup of participants, the negative predictive value of the digital stethoscope diagnosis relative to a gold standard diagnosis assigned by expert review.
Digital stethoscope Likelihood Ratio | 14 days
  Among a subgroup of participants, the likelihood ratio of the digital stethoscope diagnosis relative to a gold standard diagnosis assigned by expert review.
Digital Stethoscope diagnostic odds ratio | 14 days
  Among a subgroup of participants, the diagnostic odds ratio of the digital stethoscope diagnosis relative to a gold standard diagnosis assigned by expert review.

CONTACTS AND LOCATIONS:
Overall Officials: Eric McCollum, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Projahnnmo Research Foundation, Sylhet, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
The study will generate multiple gigabytes of de-identified individual-level data, shared as non-proprietary formats (.csv for tabular data; .wav for audio). Outcomes include treatment failure at Days 7 and 14, time to treatment failure, relapse by Day 14, modified treatment failure, outcomes stratified by age, sex, and clinic, and correct lower respiratory infection diagnosis. No participant identifiers will be shared. Metadata will include participant identification (ID) and a data dictionary. Associated documentation will include data collection instruments, methods, and final protocols. Data will be provided in formats accessible without specialized software. Common data elements, best practices, and standardized reporting approaches will be used where feasible. De-identified data, statistical analysis plans, and analytic code will be shared without restriction via public download.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Publicly shared data will be deposited into the open-source research data repository The Dataverse Project.
Access Criteria: Data will be shared by unrestricted download from The Dataverse Project open source research data repository.
URL: https://dataverse.org

REFERENCES:
- [Background] WHO. Integrated Management of Childhood Illness: Chart Booklet. 2014;https://apps.who.int/iris/bitstream/handle/10665/104772/9789241506823_Chartbook_eng.pdf.
- [Background] Ginsburg AS, Mvalo T, Nkwopara E, McCollum ED, Ndamala CB, Schmicker R, Phiri A, Lufesi N, Izadnegahdar R, May S. Placebo vs Amoxicillin for Nonsevere Fast-Breathing Pneumonia in Malawian Children Aged 2 to 59 Months: A Double-blind, Randomized Clinical Noninferiority Trial. JAMA Pediatr. 2019 Jan 1;173(1):21-28. doi: 10.1001/jamapediatrics.2018.3407. PMID 30419120
- [Background] Jehan F, Nisar I, Kerai S, Balouch B, Brown N, Rahman N, Rizvi A, Shafiq Y, Zaidi AKM. Randomized Trial of Amoxicillin for Pneumonia in Pakistan. N Engl J Med. 2020 Jul 2;383(1):24-34. doi: 10.1056/NEJMoa1911998. PMID 32609980
- [Background] McCollum ED, Park DE, Watson NL, Buck WC, Bunthi C, Devendra A, Ebruke BE, Elhilali M, Emmanouilidou D, Garcia-Prats AJ, Githinji L, Hossain L, Madhi SA, Moore DP, Mulindwa J, Olson D, Awori JO, Vandepitte WP, Verwey C, West JE, Knoll MD, O'Brien KL, Feikin DR, Hammitt LL. Listening panel agreement and characteristics of lung sounds digitally recorded from children aged 1-59 months enrolled in the Pneumonia Etiology Research for Child Health (PERCH) case-control study. BMJ Open Respir Res. 2017 Jun 30;4(1):e000193. doi: 10.1136/bmjresp-2017-000193. eCollection 2017. PMID 28883927
- [Background] Emmanouilidou D, McCollum ED, Park DE, Elhilali M. Computerized Lung Sound Screening for Pediatric Auscultation in Noisy Field Environments. IEEE Trans Biomed Eng. 2018 Jul;65(7):1564-1574. doi: 10.1109/TBME.2017.2717280. Epub 2017 Jun 19. PMID 28641244
- [Background] Hoekstra NE, Chagomerana MB, Smith ZH, Kala A, McLane I, Verwey C, Olson D, Buck WC, Mulindwa J, Gaudio A, Kapoor S, Schuh HB, Chiume M, Fitzgerald E, Elhilali M, Mvalo T, Hosseinipour M, McCollum ED. Performance of an artificial intelligence algorithm for interpreting lung sounds from children hospitalised with pneumonia in Malawi. J Glob Health. 2025 Sep 19;15:04264. doi: 10.7189/jogh.15.04264. PMID 40968644
- [Background] Kala A, Husain A, McCollum ED, Elhilali M. An objective measure of signal quality for pediatric lung auscultations. Annu Int Conf IEEE Eng Med Biol Soc. 2020 Jul;2020:772-775. doi: 10.1109/EMBC44109.2020.9176539. PMID 33018100
- [Background] Graceffo S, Husain A, Ahmed S, McCollum ED, Elhilali M. Validation of Auscultation Technologies using Objective and Clinical Comparisons. Annu Int Conf IEEE Eng Med Biol Soc. 2020 Jul;2020:992-997. doi: 10.1109/EMBC44109.2020.9176456. PMID 33018152
- [Background] Emmanouilidou D, McCollum ED, Park DE, Elhilali M. Adaptive Noise Suppression of Pediatric Lung Auscultations With Real Applications to Noisy Clinical Settings in Developing Countries. IEEE Trans Biomed Eng. 2015 Sep;62(9):2279-88. doi: 10.1109/TBME.2015.2422698. Epub 2015 Apr 13. PMID 25879837
- [Background] Park DE, Watson NL, Focht C, Feikin D, Hammitt LL, Brooks WA, Howie SRC, Kotloff KL, Levine OS, Madhi SA, Murdoch DR, O'Brien KL, Scott JAG, Thea DM, Amorninthapichet T, Awori J, Bunthi C, Ebruke B, Elhilali M, Higdon M, Hossain L, Jahan Y, Moore DP, Mulindwa J, Mwananyanda L, Naorat S, Prosperi C, Thamthitiwat S, Verwey C, Jablonski KA, Power MC, Young HA, Deloria Knoll M, McCollum ED. Digitally recorded and remotely classified lung auscultation compared with conventional stethoscope classifications among children aged 1-59 months enrolled in the Pneumonia Etiology Research for Child Health (PERCH) case-control study. BMJ Open Respir Res. 2022 May;9(1):e001144. doi: 10.1136/bmjresp-2021-001144. PMID 35577452
- [Background] Ahmed S, Sultana S, Khan AM, Islam MS, Habib GM, McLane IM, McCollum ED, Baqui AH, Cunningham S, Nair H. Digital auscultation as a diagnostic aid to detect childhood pneumonia: A systematic review. J Glob Health. 2022 Apr 23;12:04033. doi: 10.7189/jogh.12.04033. eCollection 2022. PMID 35493777
- [Background] Grzywalski T, Piecuch M, Szajek M, Breborowicz A, Hafke-Dys H, Kocinski J, Pastusiak A, Belluzzo R. Practical implementation of artificial intelligence algorithms in pulmonary auscultation examination. Eur J Pediatr. 2019 Jun;178(6):883-890. doi: 10.1007/s00431-019-03363-2. Epub 2019 Mar 29. PMID 30927097